CLINICAL TRIAL: NCT02793973
Title: The Development and Clinical Verification of Intelligent Rehabilitation System for Leg Length Discrepancy Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-01-011A
Record Dates: First submitted 2016-04-01; First posted 2016-06-08 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2016-01

CONDITIONS: Leg Length Discrepancy, Shoe Lifts
MeSH Terms: conditions — Leg Length Inequality

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 80% discrepancy lift height correction (Active Comparator): Each participant will be given 80% discrepancy shoe lift height correction through analyzing kinematic performance of center mass of body and will be required to wear the lifts in their shoes when they are walking or standing for 6 month.
  Interventions: Device: shoe lifts
- optimal lift height correction (Experimental): Each participant will be given the optimal shoe lift height correction through analyzing kinematic performance of center mass of body and will be required to wear the lifts in their shoes when they are walking or standing for 6 month.
  Interventions: Device: shoe lifts

INTERVENTIONS:
Device: shoe lifts

SUMMARY:
A structural leg length discrepancy (SLLD) is a common clinical problem. Its prevalence has been estimated at 40-70%. Those who have been suffered from limping for a long time may lead to follow-up low back pain and lower limb musculoskeletal disorders. Although lower limb triple view of x-ray is considered to be the current technique for determining LLD, it is costly and time consuming that not every hospital can afford it, and in case of radiograph, the patient is exposed to radiation. Therefore, it is necessary to develop a rapid clinical assessment method by gathering exterior parameters to build up a Regression model for measuring the discrepancy and determining LLD accurately.

While using shoe lifts to correct discrepancy is the easiest conservative intervention for LLD, there are still many controversies on how much height should be added clinically and academically. The optimal height should be added depends on feedbacks from users and gait performance. The best gait performance can be measured from kinematic performance of center mass of body during walking. Therefore, this project wants to compare treatment responses between two kinds of shoe lift height correction methods for LLD: given 80% discrepancy in shoe lift height correction through triple view of x-ray and given optimal shoe lift height correction through analyzing kinematic performance of center mass of body.

ELIGIBILITY:
Inclusion Criteria:

* aged 20 to 70
* being able to walk independently
* being diagnosed with congenital SLLD or not
* willing to cooperate to wear shoe lifts
* has smart phone and willing to record information that investigators need
* willing to sign agreement

Exclusion Criteria:

* neurological diseases (i.e. Parkinson's disease, CVA, Polio, and lower limb nerve injuries, etc.)
* diabetes along with peripheral neuropathy
* history of lower limb fracture injury or joint replacement leading to uneven leg length
* osteoporosis along with compression fracture
* foot, ankle, or knee joint deformity, osteoarthritis or soft tissue pain that disturb gait performance (ex. degenerative osteoarthritis, plantar fasciitis, and etc.)
* pregnancy
* idiopathic scoliosis
* history of psychological disease or drug addiction

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-05; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale, VAS | Changes from baseline in VAS for six month continually
  Pain fields of every participant in two groups will be recorded by APP every day for six month continually. The pain fields include：bilateral cervical, trunk, upper limb, lower limb, and foot regions, totally 10 regions.
  The score of each region is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity. The total score may range from 0-1000.

SECONDARY OUTCOMES:
Degree of comfort | Changes from baseline in comfort scale for six month continually
  Degree of comfort at foot site in two groups will be recorded by APP every day for six month continually. The score ranges from 0-10. A higher score indicates greater comfort.
areas of pain (cm^2) | Changes from baseline in areas of pain one time per week for six month
  Areas of pain in two groups will be calculated and recorded by APP. The pain fields include：bilateral cervical, trunk, upper limb, lower limb, and foot regions, totally 10 regions. The APP will give participants figures of every region. Each region will be filled with grids. Participants need to select specific grids, according to how many areas pain covers.
spatio-temporal parameters of gait | Changes from baseline in spatio-temporal parameters of gait after intervention immediately and at 4, 8, 12, 24 weeks
  GAITRite Walkway, CIR Systems, Havertown, PA, USA. The GaitRITE system was developed in response to the need for an objective way to quantify gait and ambulatory status. The GAITRite System measures spatio-temporal parameters of gait such as cadence, step length, step width, velocity, and toe-out angle, providing clinically relevant information that is useful in devising treatment plans and evaluating treatment outcomes. The system tracks parameters over time and can be used to generate progress and status reports.
three dimensional changing joint angles and trunk sway during walking | Changes from baseline in three dimensional joint angles between two segments and trunk sway during walking after intervention immediately and at 4, 8, 12, 24 week
  myoMOTION, Noraxon USA Inc., Scottsdale, AZ, USA. Wireless and portable 3D Kinematic System reveals what's unnoticeable to the naked eye, from small angular displacements to major movement pattern compensations. It contains 13 sensors fixed at bilateral dorsal side of foot, anterior medial side of tibia, lower quadrant of quadriceps, T12/L1, C7, lateral and longitudinal side of upper arm below the trapezius muscle belly, distal part of forearm and sacrum for measuring three dimensional joint angles between two segments and trunk sway during walking.
muscle activity | Changes from baseline in muscle activity after intervention immediately and at 4, 8, 12, 24 weeks
  Free EMG 300, BTS Bioengineering, Milan, Italy. BTS FREEEMG 300A is a wireless synchromyography device for dynamic muscular activity analysis. It contains eight channels for detecting muscle activity, including bilateral gluteus medius, vastus lateralis, plantar flexor, and anterior tibialis.
plantar force (kgw) | Changes from baseline in plantar force and pressure after intervention immediately and at 4, 8, 12, 24 weeks
  wireless F-Scan, Tekscan Inc., Boston, MA, USA. The F-Scan system provides dynamic pressure, force and timing information for foot function and gait analysis. Its pressure sensing film will be put between feet and shoe lifts to measureheel, medial forefoot, metatarsal head and hallux plantar force. The more even value of both sides indicates the better correction.
plantar pressure (kgw/cm^2) | Changes from baseline in plantar force and pressure after intervention immediately and at 4, 8, 12, 24 weeks
  wireless F-Scan, Tekscan Inc., Boston, MA, USA. The F-Scan system provides dynamic pressure, force and timing information for foot function and gait analysis. Its pressure sensing film will be put between feet and shoe lifts to measure heel, medial forefoot, metatarsal head and hallux plantar pressure.The more even value of both sides indicates the better correction.
contact area (cm^2) | Changes from baseline in plantar force and pressure after intervention immediately and at 4, 8, 12, 24 weeks
  wireless F-Scan, Tekscan Inc., Boston, MA, USA. The F-Scan system provides dynamic pressure, force and timing information for foot function and gait analysis. Its pressure sensing film will be put between feet and shoe lifts to measure contact area of region of interest. The value will be further calculated for determining whether the foot pronation/supination has been corrected.
Energy expenditure (Joule) | Changes from baseline in plantar force and pressure after intervention immediately and at 4, 8, 12, 24 weeks
  iPod Touch, Apple Inc., Cupertino, CA, USA. It will be fixed at lumbar-sacrum junction to measure three-dimensional instantaneous linear acceleration of center mass of body, and further to analyze kinematic performance by calculating three dimensional thrust power and thrust energy. The less energy expends, the better kinematic performance of center mass of body displays.

CONTACTS AND LOCATIONS:
Overall Officials: Si Huei Lee, Principal Investigator — Taipei Veterans General Hospital, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] DENSLOW JS, CHACE JA. Mechanical stresses in the human lumbar spine and pelvis. J Am Osteopath Assoc. 1962 May;61:705-12. No abstract available. PMID 13885486
- [Background] NELSON CR. Postural analysis and its relation to systemic disease. J Am Osteopath Assoc. 1948 Jul;47(11):555-8. No abstract available. PMID 18872347
- [Background] Greenman PE. Lift therapy: use and abuse. J Am Osteopath Assoc. 1979 Dec;79(4):238-50. No abstract available. PMID 159883
- [Background] Hoffman KS, Hoffman LL. Effects of adding sacral base leveling to osteopathic manipulative treatment of back pain: a pilot study. J Am Osteopath Assoc. 1994 Mar;94(3):217-20, 223-6. PMID 8200825
- [Background] Baylis WJ, Rzonca EC. Functional and structural limb length discrepancies: evaluation and treatment. Clin Podiatr Med Surg. 1988 Jul;5(3):509-20. PMID 3293752
- [Background] Blake RL, Ferguson HJ. Correlation between limb length discrepancy and asymmetrical rearfoot position. J Am Podiatr Med Assoc. 1993 Nov;83(11):625-33. doi: 10.7547/87507315-83-11-625. PMID 8258774
- [Background] Bhave A, Paley D, Herzenberg JE. Improvement in gait parameters after lengthening for the treatment of limb-length discrepancy. J Bone Joint Surg Am. 1999 Apr;81(4):529-34. doi: 10.2106/00004623-199904000-00010. PMID 10225798
- [Background] D'Amico JC, Dinowitz HD, Polchaninoff M. Limb length discrepancy. An electrodynographic analysis. J Am Podiatr Med Assoc. 1985 Dec;75(12):639-43. doi: 10.7547/87507315-75-12-639. No abstract available. PMID 4078719
- See also: Related Info — https://goo.gl/kwqmsn